CLINICAL TRIAL: NCT05154565
Title: The Effect of Daily Meditation on Stress, Mindfulness, Well-being, and Resilience in Student Pharmacists
Brief Title: Effect of a Daily Meditation Intervention in Student Pharmacists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Responsible Party: Principal Investigator, Spencer Harpe, Professor of Pharmacy, Midwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21029
Record Dates: First submitted 2021-09-08; First posted 2021-12-13 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Stress, Psychological; Resilience, Psychological; Mindfulness; Meditation; Well-being
Keywords: Pharmacy, Students; Education, Pharmacy
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two (2) groups. Group A is an immediate intervention group while Group B is a delayed intervention group. This allows the short-term effects of intervention to be estimated by comparing study outcomes in the treated group (Group A) with the comparison group (Group B) in Phase 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Group A) (Experimental): Meditation intervention applied during Phase 1 of the study. During Phase 2, the formal meditation intervention is not completed, but participants are followed for outcome measurement. Participants may continue to use meditation in their daily routines or return to their usual routines.
  Interventions: Behavioral: Guided meditation
- Delayed intervention (Group B) (Other): No intervention is applied in Phase 1 of the study. This group serves as the control group for Phase 1. The meditation intervention is applied in Phase 2 of the study.
  Interventions: Behavioral: Guided meditation

INTERVENTIONS:
Behavioral: Guided meditation — App-based guided meditation intervention through Headspace. This can be accessed through various mobile devices.
  Other Names: Headspace

SUMMARY:
Pharmacy school is a 3-to-4 year intensive program that demands a high level of performance from enrolled students. The fast-paced and challenging curriculum causes stress levels to rise in students. The increase in stress can negatively affect performance in the classroom, as well as affect relationships outside the classroom setting. While some level of stress may be beneficial, the substantial amount of stress experienced by pharmacy students may also negatively impact their quality of life. This proposed study aims to explore the effect a convenient intervention on perceived stress, mindfulness, well-being, and resilience as reported by student pharmacists. Headspace will be used as the main study intervention. This product is a mobile device application (aka, an app) that teaches users how to meditate through guided exercises. It contains a library of different meditation exercises the user can access from their smartphone or tablet at their own convenience. It is our hope that the use of Headspace will enhance the students' ability to practice mindfulness, which will allow them to better cope with stress in school and in future practice. This could translate into improved learning and overall well-being.

DETAILED DESCRIPTION:
This research study aims to implement a mindfulness meditation routine delivered via the smartphone application Headspace to decrease perceived stress and improve well-being, resilience, and mindfulness in student pharmacists. This product is a mobile device application (aka, an app) that teaches users how to meditate through guided exercises. It contains a library of different meditation exercises the user can access from their smartphone or tablet at their own convenience. The use of a smartphone application will allow for convenience to promote adherence with the intervention among participants. The guided meditation sessions will teach participants how to live in the present moment and handle stressful situations that may arise in the future. As a result of this program the investigators expect to see an inverse relationship between mindfulness meditation and perceived stress and direct relationships between mindfulness meditation and well-being and resilience. By learning to incorporate mindfulness meditation into their lives, participating student pharmacists may be able to develop useful tools and effectively combat overwhelming situations they may face in the future.

This study will be conducted in two phases. Participating student pharmacists will be randomly assigned to one of two groups. In Phase 1, Group A will complete four (4) weeks of guided meditation while Group B does not use the application for meditation. Changes in study outcomes will be compared from baseline to the end of the initial intervention period. In Phase 2, Group B will be complete the guided meditation intervention. Group A will continue their usual daily habits. It is possible for some students from Group A may continue to use Headspace or another similar product to continue to incorporate meditation or mindfulness into their daily routine. At the end of Phase 2, the changes in study outcomes will be examined in Group B surrounding their use of the intervention. Outcomes will also be assessed in Group A at the end of Phase 2 to examine whether there are sustained changes in study outcomes and continued usage of meditation or mindfulness practices. All participating student pharmacists will also be invited to participate in one of several focus groups sessions to discuss experiences with the use of the guided meditation application.

ELIGIBILITY:
Inclusion Criteria:

* Student pharmacists enrolled in the didactic curriculum in the Doctor of Pharmacy (PharmD) program during the Winter 2021/2022 quarter at the sponsoring institution

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in stress at 30 days | 30 days
  The change in perceived stress as measured by the Perceived Stress Scale four (4)-item measure (PSS-4; Cohen, Kamarck, & Mermelstein, 1983) will be compared between groups. This will be compared using an intent to treat approach and a per protocol approach (defined as those who were at least 80% adherent to the use of the mindfulness app). The PSS-4 yields a total score from 0 to 16 with higher scores indicating more stress.
Change from baseline in mindfulness at 30 days | 30 days
  The change in self-reported mindfulness as measured by the Five Facets of Mindfulness Questionnaire fifteen (15)-item measure (FFMQ-15; Baer, Smith, Lykins, et al., 2008) will be compared between groups. This will be compared using an intent to treat approach and a per protocol approach (defined as those who were at least 80% adherent to the use of the mindfulness app). Based on recommendations by Gu, Strauss, Crane, et al (2016), only four factors will be analyzed for change: describing, acting with awareness, non-judging, non-reactivity. Scores are derived by taking the mean response from all items and separately for each domain. Mean scores range from 1 to 5 with higher scores indicating higher levels of mindfulness.
Change from baseline in overall well-being at 30 days | 30 days
  The change in overall well-being as measured by the World Health Organization five (5)-item subjective well-being measure (WHO-5; World Health Organization, 1988) will be compared between groups. This will be compared using an intent to treat approach and a per protocol approach (defined as those who were at least 80% adherent to the use of the mindfulness app). Scores are calculated by summing the responses for each item and then multiplying by four (4). The final score ranges from 0 to 100 with higher scores indicating better well-being.
Change from baseline in resilience at 30 days | 30 days
  The change in resilience as measured by the six (6)-item Brief Resilience Scale (BRS; Smith, Dalen, Wiggins, et al., 2008) will be compared between groups. This will be compared using an intent to treat approach and a per protocol approach (defined as those who were at least 80% adherent to the use of the mindfulness app). Scores are calculated by summing the responses for each item and then dividing by six (6) to yield an overall mean score. The overall mean score ranges from 1 to 5 with higher scores indicating greater resilience.

SECONDARY OUTCOMES:
Frequency of meditation app usage | 90 days
  During the respective intervention periods, de-identified usage data provided by the application maker will be examined to identify patterns of usage by study participants. For Group A (immediate group), students will self-report their usage in Phase 2 of the study.
Acceptability of the meditation app (participant questionnaire) | 30 days
  A questionnaire was developed for this study to measure participants' opinions of the acceptability of the meditation app used. This will be administered at the end of the respective intervention period for each group (Phase 1 for Group A and Phase 2 for Group B). The questionnaire includes items on the value meditation, ease of use, and ability to incorporate the intervention into their daily schedule. Higher scores indicate more positive responses.
Continued use of meditation (participant questionnaire) | 30 days
  A questionnaire was developed for this study to measure intended use of meditation in the future. Using the theory of planned behavior as a guiding theoretical framework, the questionnaire for future use included items on intentions to practice mindfulness or meditation in the next academic quarter, attitudes towards use of mindfulness or meditation practices, subjective norms surrounding engaging in mindfulness or meditation practices, and perceived behavioral control to engage in mindfulness or meditation practices. All items are scored such that higher scores represent more positive attitudes or opinions in each area.This questionnaire will be administered at the end of the each group's respective intervention period. Higher scores indicate more positive responses.
Experience with the meditation app (participant focus group) | 120 days
  Focus group sessions will be conducted to gather feedback from participants on their experiences using meditation. Qualitative analysis will be used to construct themes identified from the participant responses.

OTHER OUTCOMES:
Change from baseline in stress at 90 days | 90 days
  In the immediate intervention group (Group A) only, the change in perceived stress as measured by the Perceived Stress Scale four (4)-item measure (PSS-4; Cohen, Kamarck, & Mermelstein, 1983) from baseline will be examined at 90 days. The PSS-4 yields a total score from 0 to 16 with higher scores indicating more stress.
Change from baseline in mindfulness at 90 days | 90 days
  In the immediate intervention group (Group A) only, the change in self-reported mindfulness as measured by the Five Facets of Mindfulness Questionnaire fifteen (15)-item measure (FFMQ-15; Baer, Smith, Lykins, et al., 2008) from baseline will be examined at 90 days. Based on recommendations by Gu, Strauss, Crane, et al (2016), only four factors will be analyzed for change: describing, acting with awareness, non-judging, non-reactivity. Scores are derived by taking the mean response from all items and separately for each domain. Mean scores range from 1 to 5 with higher scores indicating higher levels of mindfulness.
Change from baseline in overall well-being at 90 days | 90 days
  In the immediate intervention group (Group A) only, the change in overall well-being as measured by the World Health Organization five (5)-item subjective well-being measure (WHO-5; World Health Organization, 1988) will be examined at 90 days. Scores are calculated by summing the responses for each item and then multiplying by four (4). The final score ranges from 0 to 100 with higher scores indicating better well-being.
Change from baseline in resilience at 90 days | 90 days
  In the immediate intervention group (Group A) only, the change in resilience as measured by the six (6)-item Brief Resilience Scale (BRS; Smith, Dalen, Wiggins, et al., 2008) will be examined at 90 days. Scores are calculated by summing the responses for each item and then dividing by six (6) to yield an overall mean score. The overall mean score ranges from 1 to 5 with higher scores indicating greater resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Komperda, PharmD, Principal Investigator — Midwestern University; Spencer E Harpe, PharmD, PhD, Study Director — Midwestern University
Locations (1):
- Midwestern University College of Pharmacy, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Gu J, Strauss C, Crane C, Barnhofer T, Karl A, Cavanagh K, Kuyken W. Examining the factor structure of the 39-item and 15-item versions of the Five Facet Mindfulness Questionnaire before and after mindfulness-based cognitive therapy for people with recurrent depression. Psychol Assess. 2016 Jul;28(7):791-802. doi: 10.1037/pas0000263. Epub 2016 Apr 14. PMID 27078186